CLINICAL TRIAL: NCT05150522
Title: B Cell Maturation Antigen Targeted CAR-T Cells in Treatment With Relapsed and Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Principal Investigator, YuLi, Professor, Shenzhen University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEM-ONCO-012
Record Dates: First submitted 2021-11-22; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-07

CONDITIONS: Multiple Myeloma; Relapse Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA CAR-T (Experimental): BCMA CAR-T cells infusion
  Interventions: Biological: BCMA CAR-T cells

INTERVENTIONS:
Biological: BCMA CAR-T cells — BCMA CAR-T cells infusion

SUMMARY:
For the treatment of relapsed and refractory MM, the Chinese Guidelines for the Diagnosis and Treatment of Multiple Myeloma pointed out that relapsed MM is highly heterogeneous, and individualized evaluation of relapsed patients is required to determine the treatment time. Patients with biochemical recurrence with only elevated M protein do not need immediate treatment, only regular follow-up visits. For patients with CRAB manifestations or rapid biochemical relapse, treatment needs to be initiated immediately. Patients who relapse within 6 months can switch to a drug combination with other mechanisms of action; patients who relapse within 6 to 12 months should first switch to a drug combination with other mechanisms of action, or they can be retreated with the original drug; 12 months Patients with the above recurrence can use the original regimen to re-induction therapy, or switch to a drug regimen with other mechanisms of action. Bortezomib, lenalidomide, and thalidomide are currently the key drugs for the treatment of relapsed MM in China. Patients with suitable conditions should undergo autologous hematopoietic stem cell transplantation, while allogeneic hematopoietic stem cell transplantation is rarely used because of higher transplant-related mortality.

DETAILED DESCRIPTION:
For the treatment of relapsed and refractory MM, the Chinese Guidelines for the Diagnosis and Treatment of Multiple Myeloma pointed out that relapsed MM is highly heterogeneous, and individualized evaluation of relapsed patients is required to determine the treatment time. Patients with biochemical recurrence with only elevated M protein do not need immediate treatment, only regular follow-up visits. For patients with CRAB manifestations or rapid biochemical relapse, treatment needs to be initiated immediately. Patients who relapse within 6 months can switch to a drug combination with other mechanisms of action; patients who relapse within 6 to 12 months should first switch to a drug combination with other mechanisms of action, or they can be retreated with the original drug; 12 months Patients with the above recurrence can use the original regimen to re-induction therapy, or switch to a drug regimen with other mechanisms of action. Bortezomib, lenalidomide, and thalidomide are currently the key drugs for the treatment of relapsed MM in China. Patients with suitable conditions should undergo autologous hematopoietic stem cell transplantation, while allogeneic hematopoietic stem cell transplantation is rarely used because of higher transplant-related mortality.

BCMA (B cell maturation antigen), also called TNFRSF17 (TNF receptor superfamily member 17, TNF ligand superfamily member 17), is mainly expressed in plasma cells and mature B lymphocytes, is basically undetectable in other normal human cells . BCMA is the most selectively expressed receptor on the MM cell line, and its expression gradually increases with the differentiation of B cells, and it also gradually increases in the disease process of multiple myeloma. Experiments in mice found that overexpression of BCMA can induce protein kinase B, mitogen-activated protein kinase (MAPK) and nuclear factor kB (nuclear factors kB, NF-kB) signal cascade to enhance the growth and survival of MM cells, thereby Speed up the progress of MM; and down-regulation of BCMA expression can significantly reduce the formation of MM colonies and reduce the survival rate of MM cells. BCMA has become an ideal antigen target for MM because of its high selective expression in MM cell lines and its important role in normal and malignant late B cell proliferation, differentiation and antibody production.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 (≥18, ≤75) one year old, no gender limit;
2. The subject voluntarily participates in the study, and he or his legal guardian signs the "Informed Consent";
3. Definitely diagnosed as relapsed or refractory multiple myeloma: use chemotherapy regimens containing bortezomib, or chemotherapy regimens containing lenalidomide, the treatment is ineffective, or the disease progresses within 60 days after the end of the last chemotherapy;
4. The patient has one or more measurable multiple myeloma lesions, which must include any of the following:

1) Serum M protein is greater than or equal to 0.5g / dl (10g / l) 2) Urine M protein is greater than or equal to 200 mg / 24 h serum FLC ratio is abnormal 3) Serum free light chain (FLC) ≧5 mg / dL (50 mg /L) 4) Plasmacytoma that can be measured by physical examination or imaging examination 5) Myeloma cells in bone marrow ≧10% by flow cytometry or immunohistochemical examination 5. After flow cytometry or immunohistochemical examination, myeloma cells have positive BCMA expression; 6. No salvage chemotherapy was used within 4 weeks before cell therapy; 7. Within 2 weeks before cell therapy, have not received antibody drug therapy; 8. The ECOG score is 0-2 points; 9. The subject has no contraindications to peripheral blood apheresis; 10. The expected survival period is ≧12 weeks; 11. Female subjects of childbearing age must have a negative urine pregnancy test within 7 days prior to cell therapy and not during the lactation period; female or male subjects of childbearing age must take effective contraceptive measures throughout the study.

Exclusion Criteria:

1. Those who have a history of allergies to any of the ingredients in cell products;
2. The following conditions in laboratory tests: including but not limited to serum total bilirubin ≥ 1.5 mg/dl; serum ALT or AST greater than 2.5 times the upper limit of normal; blood creatinine ≥ 2.0 mg/dl; hemoglobin <80g/ l; does not rely on GCSF or other growth factors, the absolute neutrophil count is less than 1000 / mm3; no blood transfusion is required, and the platelet count is less than 30,000 / mm3;
3. According to the New York Heart Association (NYHA) cardiac function classification standards, patients with grade III or IV cardiac insufficiency; or echocardiographic examination of left ventricular ejection fraction (LVEF) <50%;
4. Abnormal lung function, blood oxygen saturation in indoor air <92%;
5. Myocardial infarction, cardiovascular angioplasty or stenting, unstable angina, or other serious clinical heart diseases within 12 months before enrollment;
6. Hypertension is grade 3 and the blood pressure is not well controlled by medication;
7. Patients with prolonged QT interval on ECG, patients with severe heart disease such as severe arrhythmia in the past;
8. Previously suffering from head injury, disturbance of consciousness, epilepsy, more serious cerebral ischemia or cerebral hemorrhage disease;
9. Need to use any anticoagulant (except aspirin);
10. Patients who need urgent treatment due to tumor progression or spinal cord compression;
11. Patients with CNS metastasis or CNS involvement symptoms (including cranial neuropathy and extensive disease or spinal cord compression);
12. The investigator determines that there are serious complications or diseases that increase the risk of the subject or affect the research, including but not limited to, for example: liver cirrhosis, recent major trauma, etc.;
13. After allogeneic hematopoietic stem cell transplantation;
14. Plasma cell leukemia;
15. Before apheresis and within 2 weeks before CAR-T cell infusion, apply more than 5 mg/d of prednisone (or an equivalent amount of other corticosteroids);
16. Patients with autoimmune diseases, immunodeficiencies or other patients who need immunosuppressive therapy;
17. There is an uncontrolled active infection;
18. Have used any CAR-T cell products or other genetically modified T cell therapies before;
19. Live vaccination within 4 weeks before enrollment;
20. HIV, HBV, HCV and TPPA/RPR infected persons, and HBV carriers;
21. The subject has a history of alcoholism, drug abuse or mental illness;
22. The subject has participated in any other clinical research within 3 months before joining this clinical research;
23. The researcher believes that the subjects have other conditions that are not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
PFS | From data of enrollment until the data of first documented progression, up to 2 years.
  Progression-Free-Survival

SECONDARY OUTCOMES:
OS | through study completion, an average of 1 year
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Li Yu, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No